CLINICAL TRIAL: NCT00750061
Title: Efficacy and Safety pf Lithium Carbonate in the Treatment of Chronic Spinal Cord Injuries: a Double-Blind, Randomized, Placebo-Controlled Clinical Trial
Brief Title: Efficacy and Safety of Lithium Carbonate in the Treatment of Chronic Spinal Cord Injuries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Spinal Cord Injury Network (Network)
Collaborators: China Rehabilitation Research Center (Other Government); Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN102A
Record Dates: First submitted 2008-08-30; First posted 2008-09-10 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo
- Lithium carbonate (Experimental): Lithium Carbonate tablet, 250mg
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — The subject start at a dosage regime of three times a day and one tablet of lithium carbonate, 250mg/table, oral administration each time for three days. The daily dose will be adjusted according to the serum lithium level and the clinical findings. Target serum lithium level is 0.6-1.2mM.
  The course of medication is 6 weeks.
  Arms: Lithium carbonate
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blinded trial. Forty patients will be randomized into two groups. The subjects in the Treatment Group will be administered with lithium carbonate, while the Control Group will receive placebo.

Each subject will receive oral lithium carbonate or placebo for six weeks. In the treatment group, the dose will be adjusted according to the serum lithium level while in the control group there will be a sham adjustment.

The outcomes will be assessed 6 weeks and 6 months after the onset of the medication. The outcomes will be compared with baseline pre-treatment data to obtain "neurological change scores." The efficacy and safety will be analyzed comparing the results of the treatment group with those of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender and 18-60 years of age;
* Subjects with chromic spinal cord injury (defined as a history of spinal cord injury for 12 months or longer);
* Subjects with ASIA - classification of A, B, or C for at least 6 months unchanged;
* Spinal cord injury vertebral level should be between C4 and T10;
* Subjects must be able to read, understand, and complete the VAS;
* Subjects who have voluntarily signed and dated an informed consent form, approved by an IRB/IEC, prior to any study specific procedures.

Exclusion Criteria:

* A history of hypersensitivity or other adverse reaction to lithium;
* Significant renal, cardiovascular, hepatic and psychiatric disease;
* Significant medical diseases or infection;
* Addison's disease;
* Debilitation or dehydration;
* Recently taken or are taking diuretics or other drugs with known interaction with lithium, such as tricyclic antidepressants, NSAIDs and tetracyclines;
* A history of alcohol abuse or drug abuse;
* Pregnant or lactating women;
* Female of childbearing potential and are unwilling to use an effective contraceptive method while enrolled in the study;
* Subjects who are currently participating in another investigational study or has been taking any investigational drug within the last 4 weeks prior to screening of this study;
* Subjects who have taken lithium for manic depression or other psychiatric conditions,and finally;
* Any criteria, which, in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mingliang Yang, MD, Ph.D, Principal Investigator — China Rehabilitation and Research Center; Tzu-Yung Chen, MD, Principal Investigator — Buddhist Tzu Chi General Hospita, Taichung Branch
Locations (2):
- China Rehabilitation and Research Center, Beijing, China
- Buddhist Tzu Chi General Hospital, Taichung Branch, Taichung, Taiwan

REFERENCES:
- [Result] Yang ML, Li JJ, So KF, Chen JY, Cheng WS, Wu J, Wang ZM, Gao F, Young W. Efficacy and safety of lithium carbonate treatment of chronic spinal cord injuries: a double-blind, randomized, placebo-controlled clinical trial. Spinal Cord. 2012 Feb;50(2):141-6. doi: 10.1038/sc.2011.126. Epub 2011 Nov 22. PMID 22105463

RESULTS

PARTICIPANT FLOW:
Groups:
- Lithium Carbonate Tablet: Lithium Carbonate: The subject start at a dosage regime of three times a day and one tablet of lithium carbonate, 250mg/table, oral administration each time for three days. The daily dose will be adjusted according to the serum lithium level and the clinical findings. Target serum lithium level is 0.6-1.2mM.
  The course of medication is 6 weeks.
Period: Overall Study
Arm/Group | Placebo | Lithium Carbonate Tablet
Started | 20 | 20
Completed | 18 | 18
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo
  Placebo: Matching placebo
- Lithium Carbonate: Lithium Carbonate
  Lithium Carbonate: The subject start at a dosage regime of three times a day and one tablet of lithium carbonate, 250mg/table, oral administration each time for three days. The daily dose will be adjusted according to the serum lithium level and the clinical findings. Target serum lithium level is 0.6-1.2mM.
  The course of medication is 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lithium Carbonate | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Year] | 38.05 (10.092) | 41.4 (6.785) | 39.624 (8.617)
Age, Customized [Number; unit: participants]
  18-30 years-old | 4 | 1 | 5
  31-40 years-old | 9 | 8 | 17
  41-50 years-old | 4 | 10 | 14
  51-60 years-old | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Changes of Neurological Scores for Baseline
Description: Changes of Motor Scores (0 ~ 100), Pin Prick Scores (0 ~ 112) and Light Touch Scores (0 ~ 112) from Baseline to Week 6 and Month 6. The higher the changes the better the functional improvement.
Time Frame: 6 months
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lithium Carbonate
Number analyzed (Participants) | 20 | 20
units on a scale
  change light touch score (wk6-d0) | -0.158 (0.688) | 0 (0)
  change light touch score (m6-d0) | 2.208 (7.141) | -0.766 (6.014)
  change pin-prick score (wk6-d0) | 0.053 (0.229) | 0.053 (0.229)
  change pin-prick score (m6-d0) | 1.906 (6.775) | -0.982 (6.498)
  change motor score (wk6-d0) | -1 (4.607) | 0 (0)
  change motor score (m6-d0) | 0.844 (6.471) | 1.316 (2.657)
Statistical Analysis 1: Comparison: Placebo vs Lithium Carbonate; change light touch score (wk6-d0); Test type: Superiority or Other; p = 0.343, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Lithium Carbonate; change light touch score (m6-d0); Test type: Superiority or Other; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Lithium Carbonate; change pin-prick score (wk6-d0); Test type: Superiority or Other; p = 1, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Lithium Carbonate; change pin-prick score (m6-d0); Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Lithium Carbonate; change motor score (wk6-d0); Test type: Superiority or Other; p = 1, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Lithium Carbonate; change motor score (m6-d0); Test type: Superiority or Other; p = 0.582, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Changes in Functional Independence Measure (FIM) Motor Subscale and Visual Analog Scale (VAS) for Pain
Description: Changes from Baseline to Week 6 and Month 6 in Functional Independence Measure (FIM) motor subscale (0 ~ 91, the higher the better), Visual Analog Scale (VAS) for pain (0 ~ 100, the less the better)
Time Frame: 6 months
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lithium Carbonate
Number analyzed (Participants) | 20 | 20
units on a scale
  change in FIM (Wk6 - D0) | 0.2 (0.4) | -0.3 (1.6)
  change in FIM (M6 - D0) | 3.5 (7.3) | 0.04 (5.4)
  change in VAS (Wk6 - D0) | 1.0 (4.0) | -9.3 (16.6)
  change in VAS (M6 - D0) | -0.9 (17.1) | -9.3 (15.3)
Statistical Analysis 1: Comparison: Placebo vs Lithium Carbonate; FIM change (Wk6 - D0); Test type: Superiority or Other; p = 0.257, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Lithium Carbonate; FIM change (M6 - D0); Test type: Superiority or Other; p = 0.168, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Lithium Carbonate; VAS change (Wk6 - D0); Test type: Superiority or Other; p = 0.013, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Lithium Carbonate; VAS change (M6 - D0); Test type: Superiority or Other; p = 0.137, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | Lithium Carbonate Tablet
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 14/20 | 16/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Lithium Carbonate Tablet (N=20)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Thirst (General disorders) | 1 (1) | 4 (4)
Pain (General disorders) | 4 (4) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Urogenital infection bacterial (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Urine output (Investigations) | 1 (1) | 0 (0)
Blood glucose abnormal (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Urine sediment present (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increase (Investigations) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 3 (4)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Self injurious behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Chromaturina (Renal and urinary disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No